CLINICAL TRIAL: NCT07017647
Title: Comparison of the Effectiveness of Conventional Treatment and Patient Education in Addition to Conventional Treatment in Individuals With Chronic Non-specific Low Back Pain: A Randomized Controlled Trial
Brief Title: Comparison of the Effectiveness of Conventional Treatment and Patient Education in Addition to Conventional Treatment in Individuals With Chronic Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Mehmet CANLI, Lecturer, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43834581758.
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-06

CONDITIONS: Low Back Pain
Keywords: Low back pain; Patient education; Conventional treatment
MeSH Terms: conditions — Low Back Pain | interventions — Conservative Treatment; Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: Randomized controlled trials
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): Conventional physiotherapy treatments will be administered to patients in the control group three days a week for six weeks. This programme will include the following treatments: electrotherapy modalities for pain relief (TENS current application), moist heat application, flexibility and strengthening exercises to stretch and strengthen the back and spinal muscles, and massage and manual therapy to relax the back muscles and reduce pain. First, TENS current will be applied for 15 minutes using an electrical stimulation device due to its pain-relieving properties. Then, moist heat application will be performed for 15 minutes. Following this, flexibility and strengthening exercises aimed at stretching and strengthening the lower back and back muscles will be performed under the supervision of a physical therapist for approximately 20 minutes. Patients will be guided to perform the exercises correctly. Thus, the total duration of the conventional physical therapy session will be 50 minut
  Interventions: Other: Conservative treatment
- Patient Education Group (Experimental): Patients in the pain education group will receive conventional physiotherapy treatments three days a week for six weeks. In addition to conventional physiotherapy treatments, patients will receive comprehensive patient education for 6 weeks. This education will be provided immediately after each conventional physiotherapy session. Patients will be asked to pay attention to and comply with the recommendations/instructions provided in this education. Comprehensive patient education includes the following: the cause of chronic back pain, negative factors that may cause discomfort and exacerbate symptoms, how to cope with back pain, ways to prevent pain, exercises and proper postures to reduce pain, and harmful movements and positions to avoid in daily life.
  Interventions: Other: Conservative treatment; Other: Patient Education

INTERVENTIONS:
Other: Conservative treatment — Conventional physiotherapy treatments will be administered to patients in both groups three days a week for six weeks. This programme will include the following treatments: electrotherapy modalities for pain relief (TENS current application), moist heat application, flexibility and strengthening exercises to stretch and strengthen the back and spinal muscles, and massage and manual therapy applications to relax the back muscles and reduce pain. First, TENS current will be applied for 15 minutes using an electrical stimulation device due to its pain-relieving properties. Then, moist heat application will be performed for 15 minutes. Following this, flexibility and strengthening exercises aimed at stretching and strengthening the lower back and back muscles will be performed under the supervision of a physical therapist for approximately 20 minutes.
Other: Patient Education — Patient education will be provided immediately after conventional physiotherapy applications in each session. Patients will be asked to pay attention to and comply with the recommendations/issues covered in this education. Comprehensive patient education includes the following: the cause of chronic back pain, negative factors that may cause discomfort and exacerbate symptoms, how to cope with back pain, ways to prevent pain, exercises and proper postures to reduce pain, and harmful movements and positions to avoid in daily life.
  Arms: Patient Education Group

SUMMARY:
Patient education is another treatment method that has recently begun to be used in patients with chronic back pain. In chronic lower back pain, factors such as the cause of the pain, negative factors that may contribute to the discomfort and exacerbate the symptoms, how to manage lower back pain, ways to prevent pain, exercises and proper postures to reduce pain, and harmful movements and positions to avoid in daily life can be included in patient education for chronic lower back pain. It has been reported that patient education in patients with chronic lower back pain can have positive effects on treatment outcomes by reducing pain, disability, and fear of movement.

DETAILED DESCRIPTION:
Low back pain is a common musculoskeletal disorder that affects approximately 80% of adults. Low back pain causes disability and functional impairment and places a significant burden on national health expenditures. Factors such as trauma, high body mass index, heavy working conditions, and weak abdominal and back muscles can cause low back pain. The most common cause of lower back pain is regional mechanical dysfunction. Rather than a single acute trauma, repetitive, cumulative traumas over time play a significant role. Risk factors such as heavy living and working conditions, poor static and dynamic posture, improper use of body mechanics, decreased strength and flexibility of abdominal and back muscles, reduced cardiovascular endurance, smoking, and vibration are known to contribute to back pain. Therefore, it is crucial to educate individuals with back pain and those at risk of developing it about these preparatory and symptom-aggravating factors. Back pain negatively affects many activities of individuals, including social life, lifting weights, carrying objects, walking, bending, standing, travelling, and dressing, thereby reducing their quality of life. Therefore, it is crucial to treat lower back pain using the effective methods recommended in the literature. If lower back pain persists for more than six months, it is classified as chronic lower back pain.

The treatment of chronic low back pain includes surgical approaches and conservative treatment. The aim of conservative treatment is to bring the patient's current condition to the best possible level. To this end, functional restoration is important in terms of both the rehabilitation of the primary damaged area and the dysfunctional secondary areas in order to accelerate the return to activity and reduce the chance of recurrence of low back pain. A treatment and rehabilitation programme is necessary to maintain the patient's optimal physiological and biomechanical fitness and to reduce the frequency of recurrent episodes of back pain. The goals of treatment in patients with chronic back pain are to reduce pain, prevent loss of condition that may develop as a result of prolonged immobilisation, prevent recurrence, resolve psychosocial problems within a multidisciplinary approach, reduce the rate of degeneration, and ensure early return to normal activities and work. In patients with chronic low back pain, pain, spasm, decreased muscle strength, and impaired posture reduce physical endurance and negatively affect the patient's functional capacity and quality of life. Conventional treatment for chronic low back pain includes conservative treatment methods. These conservative treatment methods include electrophysical agents, massage, traction, manual treatment methods, and exercise. Effective results have been reported in patients with chronic low back pain using these conservative treatment methods.

Patient education is another treatment method that has recently begun to be used in patients with chronic back pain. In chronic lower back pain, factors such as the cause of the pain, negative factors that may contribute to the discomfort and exacerbate the symptoms, how to manage lower back pain, ways to prevent pain, exercises and proper postures to reduce pain, and harmful movements and positions to avoid in daily life can be included in patient education for chronic lower back pain. It has been reported that patient education in patients with chronic lower back pain can have positive effects on treatment outcomes by reducing pain, disability, and fear of movement.

The literature highlights the limited number of studies investigating the effectiveness of patient education as an adjunct to conventional treatment in patients with chronic low back pain, suggesting that further studies in this area could make important contributions to the literature. In light of this, the aim of this study is to compare the effects of conventional treatment and patient education administered in addition to conventional treatment on pain intensity, disability status, and quality of life in patients with chronic low back pain, and to share the findings with the literature.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic low back pain by a specialist physician
* Patients who have had low back pain for more than six months
* Patients aged 18 years or older and between 18 and 65 years of age
* Patients who are not currently receiving any treatment for low back pain
* Patients with chronic non-specific low back pain

Exclusion Criteria:

* Patients with a history of surgery or trauma involving the lumbar or thoracic region,
* Patients who have received treatment for back pain in the past year,
* Patients with disc pathology, spinal fracture or dislocation, infection, malignancy, previous surgery, metabolic or inflammatory back pain, and neurological loss
* Patients who refuse to participate in the study or who do not sign the informed consent form

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-07-10 (Actual); Primary Completion 2025-11-06 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Pain Severity | 6 week
  Visual Analogue Scale (VAS) was used to determine the presence and severity of low back pain in the study participants. VAS is a practical test with high validity and reliability in pain assessment. VAS is an assessment method numbered from 0 to 10, where '0' indicates no pain and '10' indicates the presence of the most severe pain. Participants were asked to mark the degree of pain they had on this scale and recorded.

SECONDARY OUTCOMES:
Disability | 6 week
  Participants' disability level will be assessed using the Oswestry Disability Index. The Oswestry Disability Index helps to assess how low back pain affects daily living activities such as pain intensity, personal care, lifting weights, walking, sitting, standing, sleeping, sexual life, social life, and travel. Each item is scored on a scale of 0-5, with higher scores representing greater disability.
Assessment of Quality of Life | 6 week
  In assessing quality of life, the Turkish version of the SF-36 Quality of Life Assessment Scale, whose validity and reliability have been previously confirmed, will be used. The SF-36 Quality of Life Assessment Scale was developed to assess quality of life. The scale consists of a total of 36 items. A high total score on the scale indicates a high quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet CANLI, PhD., Study Director — Kirsehir Ahi Evran Universitesi
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No